CLINICAL TRIAL: NCT00142350
Title: Randomized Phase III Study of 5-FU Continuous Infusion (5-FUci) Versus CPT-11 Plus CDDP (CP) Versus S-1 Alone (S-1) in Advanced Gastric Cancer (JCOG9912)
Brief Title: A Study of 5-FUci Versus CPT-11 Plus CDDP Versus S-1 Alone in Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government); Taiho Pharmaceutical Co., Ltd. (Industry); Yakult Honsha Co., LTD (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9912; C000000062
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; 5-fluorouracil; irinotecan; cisplatin; S-1; advanced or recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: continuous infusion of 5-fluorouracil
Drug: combination of irinotecan and cisplatin
Drug: oral administration of S-1

SUMMARY:
To investigate the superiority of a combination of irinotecan and cisplatin and the non-inferiority of S-1 compared to continuous infusion of 5-FU in advanced gastric cancer

DETAILED DESCRIPTION:
From the results of our previous phase III study (JCOG9205), continuous infusion of 5-fluorouracil has remained to be a control arm of this study. This study investigates the superiority of a combination of irinotecan plus cisplatin and non-inferiority of S-1, a oral fluoropyrimidine, compared to continuous infusion of 5-fluorouracil at the point of overall survival, and the planned number of enrolled patients is 690 (230/arm).

ELIGIBILITY:
Inclusion Criteria:

1. unresectable or recurrent histologically proved gastric cancer
2. adequate oral intake
3. age 20 or older and 75 or younger
4. Performance Status (ECOG):0, 1, 2
5. measurable or unmeasurable lesions
6. preserved organ functions
7. no severe medical condition
8. no prior chemotherapy for gastric cancer
9. written informed consent

Exclusion Criteria:

1. patient with marked infection or inflammation
2. patient with severe peritoneal metastasis
3. patient with massive pleural effusion
4. patient with metastasis to CNS
5. patient with diarrhea 4 or more times per day
6. patient severe medical condition
7. patient with other concurrent malignancy affecting on survival or adverse events
8. pregnant or nursing patient or with intent to bear baby
9. patient evaluated to be inadequate by a attending doctor
10. patient requiring nutritional support

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690
Dates: Start 2000-11; Study Completion 2007-01

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
time to treatment failure
incidences of adverse events
response rate
non-hospitalized survival

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Ohtsu, MD, Study Chair — National Cancer Centr Hospital East
Locations (34):
- Japan (34):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Nagoya Medical Center, Nagoya,Naka-ku,Sannomaru,4-1-1, Aichi-ken
  - Aichi Cancer Center,Aichi Hospital, Okazaki,Kake-machi,Kuriyado,18, Aichi-ken
  - Aomori Prefectural Central Hospital, Higashitsukurimiti,2-1-1,Aomori, Aomori
  - Chiba Cancer Center Hospital, Chiba,Chuo-ku,Nitona-cho,666-2, Chiba
  - Asahi General Hospital, I-1326,Asahi, Chiba
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kyushu University Hospital, Fukuoka,Higashi-ku,Maidashi,3-1-1, Fukuoka
  - National Kyushu Cancer Center, Fukuoka,Minami-ku,Notame,3-1-1, Fukuoka
  - Federation of national public service personnel mutual aid associations Tonan Hospital, Kita 1 Nishi 6,Chuo-ku,Sapporo, Hokkaido
  - Hokkaido University Hospital, North-14 West-5 Kita-ku,Sapporo, Hokkaido
  - Hyogo Medical Center for Adults, Akashi,Kitaouji-cho,13-70, Hyōgo
  - Kobe University Graduate School of Medicine, Kobe,Chuo-ku,Kusunoki-cho,7-5-2, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun,Tomobemachi,Koibuchi,6528, Ibaraki
  - Iwate Prefectural Central Hospital, Morioka,Ueda,1-4-1, Iwate
  - Kitasato University East Hospital, Sagamihara,Asamizodai,2-1-1, Kanagawa
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Yokohama Mucipical Citizen's Hospital, Yokohama,Hodogaya-ku,Okazawa-cho,56, Kanagawa
  - Yokohama City University Medical Center, Yokohama,Minami-ku,Urafunecho,4-57, Kanagawa
  - Kochi Health Science Center, Kochi,Ike,2125-1, Kochi
  - Kumamoto Regional Medical Center Hospital, Kumamoto,Honjo,5-16-10, Kumamoto
  - Kyoto University Hospital, Kyoto,Sakyo-ku,Syogoinkawara,54, Kyoto
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Saku Central Hospital, Saku,Usuda,197, Nagano
  - Osaka Medical College, Takatsuki,Daigakucho,2-7, Osaka
  - Saitama Medical School Hospital, Iruma-gun,Moroyama-machi,Morohongo,38, Saitama
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - Div. of Gastrointestinal Oncology, Shizuoka Cancer Center, Sunto-gun, Nagaizumi-cho, Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - Showa University School of Medicine, Shinagawa-ku,Hatanodai,1-5-8, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- [Derived] Kurokawa Y, Boku N, Yamaguchi T, Ohtsu A, Mizusawa J, Nakamura K, Fukuda H. Inter-institutional heterogeneity in outcomes of chemotherapy for metastatic gastric cancer: correlative study in the JCOG9912 phase III trial. ESMO Open. 2016 Feb 8;1(1):e000031. doi: 10.1136/esmoopen-2015-000031. eCollection 2016. PMID 27843586
- [Derived] Takahari D, Boku N, Mizusawa J, Takashima A, Yamada Y, Yoshino T, Yamazaki K, Koizumi W, Fukase K, Yamaguchi K, Goto M, Nishina T, Tamura T, Tsuji A, Ohtsu A. Determination of prognostic factors in Japanese patients with advanced gastric cancer using the data from a randomized controlled trial, Japan clinical oncology group 9912. Oncologist. 2014 Apr;19(4):358-66. doi: 10.1634/theoncologist.2013-0306. Epub 2014 Mar 25. PMID 24668328
- [Derived] Boku N, Yamamoto S, Fukuda H, Shirao K, Doi T, Sawaki A, Koizumi W, Saito H, Yamaguchi K, Takiuchi H, Nasu J, Ohtsu A; Gastrointestinal Oncology Study Group of the Japan Clinical Oncology Group. Fluorouracil versus combination of irinotecan plus cisplatin versus S-1 in metastatic gastric cancer: a randomised phase 3 study. Lancet Oncol. 2009 Nov;10(11):1063-9. doi: 10.1016/S1470-2045(09)70259-1. Epub 2009 Oct 7. PMID 19818685
- See also: Related Info — http://www.jcog.jp/